CLINICAL TRIAL: NCT03679637
Title: The Feasibility, Usability and Acceptability of a Tablet-based Aphasia Therapy in the Acute Phase After Stroke
Brief Title: Tablet-based Aphasia Therapy in the Acute Phase After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Neurologie, Principal Investigator, clinical professor Veerle De Herdt, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2018/1006
Record Dates: First submitted 2018-09-07; First posted 2018-09-20 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Aphasia; Stroke, Acute
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Each participant will receive a tablet-based aphasia therapy
  Interventions: Behavioral: Tablet-based aphasia therapy

INTERVENTIONS:
Behavioral: Tablet-based aphasia therapy — patients will independently practice with a speech app during hospitalisation

SUMMARY:
As aphasia is one of the most common and disabling disorders following stroke, in many cases resolving in long-term deficits, it is now thought that intensive aphasia therapy is effective, even in the chronic phase following stroke. However, as intensive aphasia rehabilitation is difficult to achieve in clinical practice, tablet-based aphasia therapies are explored to further facilitate language recovery. Although there is mounting evidence that computer-based treatments are effective, it is also important to assess the feasibility, usability and acceptability of these technologies, especially in the acute phase post stroke. The investigators assume that tablet-based aphasia therapy is a feasible treatment option for patients with aphasia in the acute phase following stroke. The researchers also believe that the specific app that will be used in therapy is user-friendly and that it will be well accepted by this specific patient population.

DETAILED DESCRIPTION:
The study is a prospective study, with each participant undergoing testing approximately within three days after inclusion in the study (immediately prior to tablet-based aphasia therapy). Based on the results of diagnostic testing (standard of care in the acute phase), therapy will be tailored for each individual. After two short training sessions, patients will independently practice with the app during hospitalisation, guided by a user-friendly instruction sheet. Patients will be encouraged to practice as much as possible, with a minimum of 30 minutes per day. Exercises will be selected by the speech-language therapist based on diagnostic results and will be adjusted for difficulty and type of exercise during treatment based on performance rates. the aim of the study is to investigate the feasibility, usability and acceptability of a tablet-based aphasia therapy in patients with aphasia in the acute phase following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with aphasia after an ischemic or hemorrhagic stroke
* Maximum 2 weeks post-stroke
* Minimum 18 years old
* A minimum proficient language level of Dutch
* Imaging (CT or MRI) prior to inclusion
* Signed informed consent

Exclusion Criteria:

* Presence of severe psychiatric disorders and/or cognitive disorders that hinder the use of the tablet-based aphasia therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of a tablet-based aphasia therapy via the recruitment rate | from date of inclusion to date of hospital discharge, assessed up to 20 weeks
  Recruitment rate: number of patients enrolled versus total patients meeting study criteria + notation of reasons why patients did not enroll
Feasibility of a tablet-based aphasia therapy via the retention rate | from date of inclusion to date of hospital discharge, assessed up to 20 weeks
  Retention rate: number of patients continuing to use the mobile tablet until the time of discharge + notation of reasons why patients did not continue practicing
Feasibility of a tablet-based aphasia therapy via the adherence rate, | from date of inclusion to date of hospital discharge, assessed up to 20 weeks
  Adherence rate: time patients practiced versus time advised to practice + notation of reasons why patients did not practice the advised time
Feasibility of a tablet-based aphasia therapy via protocol deviations | from date of inclusion to date of hospital discharge, assessed up to 20 weeks
  Notation of any protocol deviations
Usability of a tablet-based aphasia therapy via a self-prepared usability questionnaire, | date of hospital discharge, an average of 1 week
  Self-prepared usability questionnaire: patients will need to fill in a 5 question survey (5-point Likert scale) measuring the usability of a tablet-based therapy. Minimum score is 1 (= totally not agree), maximum score is 5 (= totally agree)
Usability of a tablet-based aphasia therapy via an observational checklist | date of hospital discharge, assessed up to 20 weeks
  Self-prepared observational checklist: patients will be observed during a therapy session. Different sub-tasks will be scored for independency on a 3-point scale. Minimum score is 1 (completely dependent), maximum score is 3 (= completely independent)
Usability of a tablet-based aphasia therapy via within-task improvements of the app | from date of inclusion to date of hospital discharge, assessed up to 20 weeks
  Notation of exercises performed with the app
Acceptability of a tablet-based aphasia therapy via a vertical VAS-scale for satisfaction | date of hospital discharge, an average of 1 week
  Vertical visual anologue scale (VAS) for satisfaction: patients have to indicate their general level of satisfaction post-intervention on a vertical VAS-scale. Minimum score is 0 (= not satisfied), maximum score is 100 (= very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Veerle De Herdt, Principal Investigator — University Ghent
Locations (1):
- University Hospital, department of neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Cock E, Batens K, Feiken J, Hemelsoet D, Oostra K, De Herdt V. The feasibility, usability and acceptability of a tablet-based aphasia therapy in the acute phase following stroke. J Commun Disord. 2021 Jan-Feb;89:106070. doi: 10.1016/j.jcomdis.2020.106070. Epub 2020 Dec 29. PMID 33418143